CLINICAL TRIAL: NCT04596241
Title: Effect of BTL-899 Device for Non-invasive Lipolysis and Improvement of Muscle Tone in Upper Arms
Brief Title: Non-invasive Lipolysis and Improvement of Muscle Tone in Upper Arms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-899_100
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Fat Disorder
MeSH Terms: conditions — Lipid Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental (Experimental): Subjects will be required to complete four (4) treatment visits and two follow-up visits. All of the study subjects will receive the treatment with the subject device.
  Interventions: Device: BTL-899

INTERVENTIONS:
Device: BTL-899 — Treatment with intensities of a magnetic field and radiofrequency energy just below the patient's tolerance threshold.

SUMMARY:
This study will evaluate the clinical efficacy and safety of the BTL-899 device for changes in subcutaneous fat tissue and muscle tissue of arms. The study is a prospective multi-center open-label single-arm study. The subjects will be enrolled and assigned into a single study group. Subjects will be required to complete four (4) treatment visits and two follow-up visits. All of the study subjects will receive the treatment with the subject device.

DETAILED DESCRIPTION:
This study will evaluate the clinical efficacy and safety of the BTL-899 device for changes in subcutaneous fat tissue and muscle tissue of arms. The study is a prospective multi-center open-label single-arm study. The subjects will be enrolled and assigned into a single study group. Subjects will be required to complete four (4) treatment visits and two follow-up visits. All of the study subjects will receive the treatment with the subject device.

At the baseline visit, MRI imaging will be performed; the subject's weight and arm circumference will be recorded. Photos of the treated area will be taken.

The treatment administration phase will consist of four (4) treatments, delivered 5-10 days apart. The applicator of BTL-899 will be applied over the treatment area. The device will induce visible muscle contractions along with heating of the subcutaneous fat. Each therapy session will last 30 minutes.

At the last therapy visit, the subject's weight and arm circumference will be recorded, and photos of the treated area will be taken. In addition, subjects will receive a Subject Satisfaction Questionnaire to fill in.

Safety measures will include documentation of adverse events (AE), including the subject's experience of pain or discomfort after each procedure. Following each treatment administration and at all of the follow-up visits, subjects will be checked for immediate post-procedure adverse event assessment.

During the post-procedure visits (at 1-month and 3-month follow-up visits), the subjects will undergo a MRI imaging. Also, the subject's satisfaction will be noted, and weight with arm circumference will be recorded. Photographs of the treated area will be taken. In addition, subjects will receive a Lifestyle Change Questionnaire to fill in.

ELIGIBILITY:
Inclusion Criteria:

* Arm fat layer > 1.0 cm
* Age > 21 years
* Voluntarily signed an informed consent form
* BMI ≤ 35 kg/m2
* Women of child-bearing potential are required to use birth control measures during the
* whole duration of the study
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring during study participation
* Subjects willing and able to maintain her regular (pre-procedure) diet and exercise regimen without affecting significant change in either direction during study participation

Exclusion Criteria:

* Electronic implants (such as cardiac pacemakers, defibrillators, and neurostimulators)
* Metal implants
* Drug pumps
* Malignant tumor
* Pulmonary insufficiency
* Injured or otherwise impaired muscles
* Cardiovascular diseases
* Disturbance of temperature or pain perception
* Hemorrhagic conditions
* Septic conditions and empyema
* Acute inflammations
* Systemic or local infection such as osteomyelitis and tuberculosis
* Contagious skin disease
* Elevated body temperature
* Pregnancy, postpartum period, nursing, and menstruation
* Intrauterine device (IUD)
* Swollen or neoplastic tissues, space-occupying lesions or skin eruptions in the treatment area
* Basedow's disease

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
The evaluation of structural changes of subcutaneous tissues of the of the upper arms | 4 months
  The evaluation of structural changes of subcutaneous tissues between pre-treatment and post-treatment based on MRI imaging through measurements of the thickness of subcutaneous tissues
The evaluation of structural changes of subcutaneous tissues of the of the upper arms | 4 months
  The evaluation of structural changes of subcutaneous tissues between pre-treatment and post-treatment based on MRI imaging through evaluation of tissue composition and morphology.
The evaluation of change in adipose layer thickness | 4 months
  The evaluation of change in adipose layer thickness between pre-treatment and post-treatment based on arm circumference measurements.

SECONDARY OUTCOMES:
Patient's satisfaction with study treatment measured via questionnaires | 4 months
  To determine the patient's satisfaction with study treatment for non-invasive lipolysis and improvement of muscle tone in upper arms. The 5-point Likert scale Satisfaction questionnaire will be used to evaluate the participant's satisfaction with the therapy outcome. Subject satisfaction will be assessed after the last therapy visit and during the follow-up visits with 4-therapy related questions with answer "Strongly agree" will be the best possible answer and "Strongly disagree" the worst.
Evaluation of the Therapy's Safety Measured Via Therapy Comfort Questionnaire | 4 months
  The outcome will further be measured through the occurrence of adverse events or lack thereof. On Numerical Analog Scale (0-10), where 0 represents 'no pain' and 10 represents 'worst possible pain' select the level of pain experienced during the treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Chicago Cosmetic Surgery and Dermatology, Chicago, Illinois
  - Maryland Laser Skin and Vein Institute, Hunt Valley, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacob C, Weiss RA. Simultaneous HIFEM and Synchronized RF Procedure Can Be Effectively Used for Increasing Muscle Mass and Decreasing Fat in the Upper Arm. J Clin Aesthet Dermatol. 2023 Feb;16(2):50-54. PMID 36909865